CLINICAL TRIAL: NCT05672836
Title: A Randomized, Double-Blind, Placebo-controlled Trial to Evaluate Efficacy and Safety of a Novel Sodium-Glucose Cotransporter 2 Inhibitor, Enavogliflozin Compared to Placebo on Reducing Major Cardiovascular Events or Worsening Heart Failure in Patients With Severe Aortic Stenosis Who Underwent Transcatheter Aortic Valve Replacement (TAVR) and With Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: ENAVOgliflozin Outcome Trial in Patients With Severe Aortic Stenosis After Transcatheter Aortic Valve Replacement
Acronym: ENAVO-TAVR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Professor, Cardiology, Asan Medical Center Heart Institute, Valvular Heart Disease Center, Ischemic Heart Disease Center, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMCCV2023-01
Record Dates: First submitted 2023-01-01; First posted 2023-01-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis; Heart Failure
Keywords: Transcatheter Aortic Valve Implantation; heart failure with preserved ejection fraction; Sodium-glucose cotransporter-2 inhibitor; transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Failure | interventions — Enavogliflozin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enavogliflozin Group (Experimental): 0.3 mg 1 tablet once daily
  Interventions: Drug: Enavogliflozin
- placebo as add-on to standard of care treatment group (Placebo Comparator): Placebo matching enavogliflozin
  Interventions: Drug: Standard-of-Care

INTERVENTIONS:
Drug: Enavogliflozin — 0.3 mg 1 tablet once daily
  Arms: Enavogliflozin Group
Drug: Standard-of-Care — Standard-of-Care medical therapy plus Enavogliflozin matching placebo
  Other Names: Standard-of-Care medical therapy
  Arms: placebo as add-on to standard of care treatment group

SUMMARY:
The goal of this trial is to to determine whether use of a novel SGLT2 inhibitor, Enavogliflozin 0.3 mg once daily is superior to placebo, when added to standard-of-care, in reducing the composite of major cardiovascular events and Heart Failure events (hospitalization for Heart Failure or urgent Heart Failure visit) among patients who underwent transcatheter aortic valve replacement for severe aortic stenosis and with heart failure with preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥19 with symptomatic aortic stenosis who underwent successful transcatheter aortic valve replacement (TAVR)* (either native valve or valve in valve with any approved/marketed device).

* A successful TAVI is defined as device success according to the VARC-2(Valve Academic Research Consortium 2) and VARC-3 criteria:

1. correct positioning of a single prosthetic heart valve into the proper anatomical location AND
2. intended performance of the prosthetic heart valve (mean aortic valve gradient <20 mmHg, peak velocity <3 m/s, no moderate or severe prosthetic valve regurgitation) AND
3. absence of periprocedural complications (any type of stroke, life-threatening bleeding, acute coronary artery obstruction requiring intervention, major vascular complication requiring intervention, unresolved acute valve thrombosis, or any requirement of a repeat procedure).

2. Heart Failure with Mildly Reduced or Preserved Ejection Fraction

1. Left ventricular ejection fraction (LVEF) ≥40%
2. structural heart disease_Left ventricular hypertrophy (LVH) or Left atrial enlargement

   A. Left ventricular hypertrophy (LVH) with septal thickness or posterior wall thickness ≥ 1.1 cm or

   B. Left atrial (LA) enlargement with at least one of the following: LA width (diameter) ≥3.8 cm or LA length ≥ 5.0 cm, or LA area ≥ 20cm2, or LA volume ≥ 55mL or LA volume index ≥ 29mL/m.
3. NT-proBNP ≥ 300 pg/mL (for patients without ongoing atrial fibrillation) or NT-proBNP must be ≥ 600 pg/mL (for patients with ongoing atrial fibrillation).

3. Patients who voluntarily participated in the written agreement

Exclusion Criteria:

1. Acute decompensated Heart Failure (exacerbation of chronic Heart Failure) requiring intravenous diuretics, vasodilators, inotropic agents, or mechanical support, or hemodynamic instability following the transcatheter aortic valve replacement procedure.
2. Currently receiving therapy with an SGLT2 inhibitor within 4 weeks prior to randomization; discontinuation of current use of SGLT2 inhibitor for the purposes of study enrolment is not permitted.
3. Known allergy, hypersensitivity, or previous intolerance to an SGLT2 inhibitors.
4. HF with reduced ejection fraction (LVEF <40%).
5. Type 1 diabetes mellitus or diabetes ketoacidosis.
6. Chronic cystitis and/or recurrent urinary tract infection (≥2 times within 1 year).
7. Stroke or transient ischemic attack within 12 weeks prior to enrollment.
8. Symptomatic persistent hypotension and/or a systolic blood pressure (SBP) < 95 mm Hg at screening or at randomization.
9. SBP ≥180 mmHg irrespective of treatment or SBP ≥160 mmHg with at least ≥3 antihypertensive drugs at screening or randomization.
10. Heart failure due to any of the following causes; known infiltrative cardiomyopathy (e.g. amyloid, sarcoid, lymphoma, endomyocardial fibrosis, haemochromatosis, Fabry disease), active myocarditis, constrictive pericarditis, cardiac tamponade, known hypertrophic obstructive cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy/dysplasia (ARVD), or uncorrected primary valvular disease.
11. Severe renal insufficiency (eGFR <30 ml/min/1.73 m2 of body-surface area based on the Modification of Diet in Renal Disease (MDRD) formula) or end-stage renal disease or requiring dialysis at the time of screening.
12. Acute or chronic liver disease with severe impairment of liver function (e.g., ascites, esophageal varices, coagulopathy) or serum levels of transminases or alkaline phosphatase more than two times the upper limit of normal at screening.
13. Chronic pulmonary disease requiring home oxygen, oral steroid therapy or hospitalization for exacerbation within 12 months, or significant chronic pulmonary disease in the Investigator's opinion, or primary pulmonary arterial hypertension.
14. Current or suspicious malignancy or history of malignancy within 5 years
15. Uncontrolled anaemia or haemoglobin <9g/dl
16. Uncontrolled hypothyroidism or arrhythmia or tachycardia
17. Current ongoing alcoholic or drug addict
18. Subjects with non-cardiac co-morbidities with life expectancy less than 12 months
19. Planned major high-risk operation after transcatheter aortic valve replacement (TAVR)
20. Women of childbearing age who have not reached a consensus on the use of highly effective contraception. Pregnancy or breastfeeding.
21. Participation in other clinical trials, However, where at least one or more conditions are satisfied, it could be an exception according to an investigator's discretion;

    * Participating in the observational study expected no effect on the safety and/or effectiveness evaluation of this trial.
    * Screening failed before any interventional factor is involved.
    * Participants who have completed their involvement in clinical trials and have surpassed a 4-week period since their last administration of the investigational drug.
    * Participated in academic trials like strategic or medical device comparison studies conducted under standard therapy provided that there is no additional risk or a specific procedure to a subject and no interference between this trial and other studies.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to first occurrence of a composite of major adverse cardiovascular events* or hospitalization for heart failure | 12 months
  Time from randomization to the first occurrence of a composite of major adverse cardiovascular events* or hospitalization for heart failure at 12 months after randomization.
  *Major adverse cardiovascular events included death from any causes, nonfatal myocardial infarction, or nonfatal stroke.
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event is considered to have occurred if any one of several different events is observed.

SECONDARY OUTCOMES:
Event rate of death from any cause | 12 months
Event rate of nonfatal myocardial infarction | 12 months
Event rate of nonfatal stroke | 12 months
Event rate of hospitalization for heart failure | 12 months
Event rate of Composite renal endpoint | 12 months
  Composite renal endpoint, defined as time to first occurrence of (1) chronic dialysis; (2) renal transplantation; (3) sustained reduction of ≥40% in estimated glomerular filtration rate (GFR); or (4) sustained estimated GFR <15 mL/min/1.73 m2 for patients with baseline estimated GFR ≥30 mL/min/1.73 m2.
Event rate of Rehospitalization for any reason | 12 months
Changes in measures of cardiac volume and function assessed by serial echocardiography | 12 months
  left ventricular ejection fraction(LVEF), LV end-diastolic volume index (LVEDVI), LV end-systolic volume index (LVESVI), left atrial volume index (LAVI), and the ratio of early transmitral Doppler velocity/early diastolic annular velocity (E/e')
Changes in New York Heart Association (NYHA) functional class and the Kansas City Cardiomyopathy Questionnaire (KCCQ) summary score | 12 months
  New York Heart Association (NYHA) Functional Classification on a scale from I to IV, with higher scores indicating severe symptoms and physical limitations associated with heart failure.
  the Kansas City Cardiomyopathy Questionnaire (KCCQ)on a scale from 0 to 100, with higher scores indicating fewer symptoms and physical limitations associated with heart failure.
Serial change in NT-proBNP | 12 months
  N-terminal (NT)-pro hormone BNP (NT-proBNP)
Event rate of the safety events | 12 months
  The safety events are defined as;
  * Serious adverse events
  * Adverse events leading to treatment discontinuation
  * Adverse events of special interest(AESI)
    * Hypoglycemia, genitourinary infections, hepatic injury, decreased renal function, ketoacidosis, events leading to lower limb amputation
  * AESIs leading to treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Seung-jung Park, MD, Study Chair — Professor, Cardiology, Asan Medical Center Heart Institute, Valvular Heart Disease Center, Ischemic Heart Disease Center
Locations (31):
- South Korea (31):
  - Bucheon Sejong Hospital, Bucheon-si
  - Gyeongsang National University Changwon Hospital, Changwon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Incheon Sejong Hospital, Incheon
  - Inha University Hospital, Incheon
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Dong-A Medical Center, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Seoul university Bundang hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - SNU Boramae Medical Center, Seoul
  - The Catholic Univ. of Korea Eunpyeong St. Mary's hospital, Seoul
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon
  - Uijeongbu Eulji Medical Center, Eulji University, Uijeongbu-si
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Undecided